CLINICAL TRIAL: NCT06425692
Title: Enhancing Palliative Care in ICU (EPIC) - Work Package 3
Brief Title: Work Package 3 Education for ICU Clinicians in Basic Palliative Care
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2023-2676
Record Dates: First submitted 2024-05-01; First posted 2024-05-22 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: ICU; Staff Attitude; Learning; Palliative Care, Patient Care
Keywords: multi-center study; ICU staff; EU-Horizon
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Education on basic palliative care (Other): Blended learning for ICU staff and online webinars. The aim is to teach the basics of palliative care on a cognitive, affective and psychomotor level.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Education on basic palliative care via e-learning + webinar to deepen knowledge.

SUMMARY:
The EPIC project aims at sustainably improving palliative care for seriously ill patients and their families in ICUs. To this aim, an interdisciplinary consortium is working together to provide a new practical palliative care model using telemedicine. The project is the first European intervention study on palliative care in the ICU using a systems- based approach with proactive patient identification, checklist and blended learning designed to meet the specific needs of ICU staff.

EPIC's vision is to contribute to a change in awareness from a narrow focus on prolonging life to a more holistic approach to care.

The development of blended learning for intensive care staff is the task of Work Package (WP) 3. The aim is to improve the attitude, understanding and self-confidence of ICU staff. Blended learning is to be developed and implemented for this purpose. The aim is to teach the basics of palliative care on a cognitive, affective and psychomotor level.

Due to the international character of the project, it is to be developed in English with subtitles in the local languages. In addition a workshop with patient and family advisors will be conducted.

DETAILED DESCRIPTION:
Background Around 10% of all deceased people in the population die after being admitted to an intensive care unit (ICU). These patients may have distressing symptoms and may receive more intensive life-prolonging treatment than they would have chosen themselves. This can lead to family stress, but also to mental distress among intensive care staff.

The EPIC project aims at sustainably improving palliative care for seriously ill patients and their families in ICUs. To this aim, an interdisciplinary consortium is working together to provide a new practical palliative care model using telemedicine. The project is the first European intervention study on palliative care in the ICU using a systems-based approach with proactive patient identification, checklist and blended learning designed to meet the specific needs of ICU staff. EPIC's vision is to contribute to a change in awareness from a narrow focus on prolonging life to a more holistic approach of care.

Objectives of Work Package (WP) 3 The aim is to improve the attitude, understanding and self-confidence of ICU-staff. Blended learning will be developed and implemented for this purpose. The aim is to teach the basics of palliative care on a cognitive, affective and psychomotor level. Due to the international character of the project, it is to be developed in English with subtitles in the local languages. In addition a workshop with patient and family advisors should conducted.

Development and implementation of blended learning

The blended learning program is to be completed by all ICU staff participating in the study during the crossover period of 4 weeks prior to the intervention. The curriculum will be developed in close collaboration with another work package. The main aim is to teach the standardized EPIC procedures using the following questions:

1. Why is palliative care necessary?
2. When to call for a specialist palliative care consultation?
3. How to message palliative care?
4. What are the critical elements of palliative care in the ICU?

Participants first complete the eLearning programme. This is made available to them via the data-secured open-source platform: BeST, Charite. Participants will then take part in interactive online workshops moderated by the investigators involved in the study. The workshop curriculum also focuses on communication skills training and open questions after the eLearning. Two workshops of 90 minutes each will be offered to allow all ICU staff to participate. In addition, a pocket card for symptom assessment, communication and care planning will be developed and handed out at each workshop.

Evaluation of the impact of the training The evaluation of blended learning takes place at different times. On one hand, the validated CPD Response Questionnaire, a 12-item questionnaire to assess the impact of CPD activities on changes in clinical behavioral intentions, will be used. CPD activities can be used as a way of indicating that new knowledge can lead to changes in practice.

Which changes the investigators want to measure will become apparent during the development of the curriculum.

The comparative self-assessment (CSA) gain is used to evaluate the specific learning effects in relation to the increase in knowledge, attitudes and skills. Here, the participants assess their own increase in knowledge in the post/this assessment. The information is assessed using German school grades (1 = very good, 6 = unsatisfactory). Subsequently, the learning gain on the levels of attitude and knowledge can be calculated as CSA Gain [%] = ((MWpre-MWpost)/(Mwpre-1)) x 100.

The learning objectives will be based on the curriculum to be developed, so the questionnaire will also be submitted as an amendment. Both questionnaires will be made available to participants via a link and/or QR code using SoSci Survey tool. The CPD is to be surveyed before and after blended learning and after six months, and the CSA gain after blended learning and also after six months.

The questionnaires are available in English and will be translated back and forth according to the state of the art. Reminders for the follow-up questionnaires will be sent to the participants by e-mail. Results will be communicated to the investigators at other sites and used to update the curriculum after the intervention study has ended.

Conducting and evaluation of the patients and family workshop A co-workshop will be held with patients and relatives to integrate their perspectives and needs in terms of skills and knowledge of professional caregivers. This will then also be evaluated, whereby the content to be developed will provide the items of the evaluation. The evaluation is also collected as an online questionnaire via SoSci.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years
* ICU staff and participants of the EPIC intervention study (physician, nurse)
* participants of patients and family workshops
* agreement to participate in the study

Exclusion Criteria:

* <18 years
* rejection of study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
CSA-gain | e-Learning: 45 minutes, CSA-gain immediately after e-learning and 6 months post e-learning.
  The comparative self-assessment (CSA) gain is used to evaluate the specific learning effects in relation to the increase in knowledge, attitudes and skills [2]. Here, the participants assess their own increase in knowledge in the post/this assessment. The information is assessed using german school grades (1 = very good, 6 = unsatisfactory). Subsequently, the learning gain on the levels of attitude and knowledge can be calculated as "Comparative Self-Assessment Gain" (CSA Gain [%] = ((MWpre- MWpost)/(Mwpre-1)) x 100) using specific outcome evaluation.
CPD Response Questionnaire ("Continuing professional development") | Right before starting the 45-minute e-learning session + immediately after the completion of one of the offered online workshops (to be held on two Thursdays per month for 5 years) + 6 months post blended learning.
  12-item questionnaire to assess the impact of CPD activities on changes in clinical behavioural intentions

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Raupach T, Munscher C, Beissbarth T, Burckhardt G, Pukrop T. Towards outcome-based programme evaluation: using student comparative self-assessments to determine teaching effectiveness. Med Teach. 2011;33(8):e446-53. doi: 10.3109/0142159X.2011.586751. PMID 21774642
- [Background] Legare F, Freitas A, Turcotte S, Borduas F, Jacques A, Luconi F, Godin G, Boucher A, Sargeant J, Labrecque M. Responsiveness of a simple tool for assessing change in behavioral intention after continuing professional development activities. PLoS One. 2017 May 1;12(5):e0176678. doi: 10.1371/journal.pone.0176678. eCollection 2017. PMID 28459836